CLINICAL TRIAL: NCT07031024
Title: Tabacco Cessation: Evaluation of Patient Perceptions and Professional Practices in the Odontology Department of the Nice Institute of Oral Medicine
Brief Title: Tabacco Cessation in Hospital Services
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Odonto01
Record Dates: First submitted 2025-03-21; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Survey on smokers , feelings and perception of tabacco cessation , delivery by a dentist
- Hospital practitioner: Survey on hospital dentists, knowledge, attitude, and practice

SUMMARY:
Tobacco poses a health risk, whatever the method of consumption. According to the baro cancer 2021 : Only 23% of smokers say they have discussed smoking with a healthcare professional in the last 12 months. Studies in France on the practitioner's point of view have mainly been carried out in private practice, and at least 2 years ago. Few studies have looked at the patient's point of view. To date, no studies have been carried out in France on the patient's point of view. This is why the aim of our study is to: current state of smoking cessation in a hospital services: knowledge, attitudes and practices, from the point of view of the practitioner and the patient. Evaluation via a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Female male non gendered.
* Over 18 years old
* Whatever their state of healthRegular smoker: According to the Institut national de prévention et d'éducation pour la santé (INPES), a regular smoker is someone who reports smoking at least one cigarette (or equivalent) a day.
* Whether or not they use any other form of 'drug'.
* Whatever the reason for their consultation.
* Signature of no objection form
* Praticiens:- Male , Female non gendered
* Age 18 years
* General practitioner at CHU ( Professor - MCU - Assistant - Associate)
* Specialist at the University Hospital (Professor - MCU - Assistant - Associate)
* Intern (oral medicine - oral surgery - orthodontics)
* student (4th, 5th and 6th year)"

Exclusion Criteria:

* Patients: Ex-smoker patients
* Non-smokers
* Patients under guardianship
* Patients with language difficulties
* Praticiens: - Non-dentistry students
* Student in dentistry without clinical practice (2nd, 3rd year)
* Practitioner with exclusive private practice"

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Smoking patients attending the Nice Institute of Oral Medicine. Practitioners, interns and 4th, 5th and 6th year students.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Description of the participant's group | At the inclusion
  Participant's questionnaire: 16 questions without score

SECONDARY OUTCOMES:
Identify the factors that influence responses to questions (Demographic characteristics) | At the inclusion
  Demographic characteristics of participants: gender and age.
Identify the factors that influence responses to questions (the knowledge particiapnts) | At the inclusion
  Questionnaire:the knowledge participants without score
Identify the factors that influence responses to questions (patients prejudices) | At the inclusion
  Questionnaire:the patients prejudices without score
Identify the factors that influence responses to questions ( Practionner status) | At the inclusion
  Questionnaire: Professionnal status of practionners without score

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France